CLINICAL TRIAL: NCT01334489
Title: Arabin Cervical Pessary for Prevention of Preterm Birth in Cases of Twin-to-twin Transfusion Syndrome Treated by Fetoscopic Laser Coagulation: The PECEP Laser Trial
Brief Title: The Trial of Pessary After Laser for TTTS
Acronym: PECEPLASER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis unfavorable to continue the study
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Maternal-Infantil Vall d´Hebron Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Bürgerhospital Frankfurt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PECEP_LASER Trial
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Premature Birth
Keywords: Monochorionic pregnancy; Twin to twin transfusion syndrome; Cervical pessary; Cervical length
MeSH Terms: conditions — Premature Birth; Fetofetal Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual management (No Intervention): Usual management of monochorionic pregnancy without the pessary placement
- Arabin Cervical Pessary (Other): The pessary will be inserted 24 hours after fetal surgery in the exploration room. This procedure does not need anaesthesia and it does not need to be done in a surgery room. During the following explorations the correct placement of the pessary is assessed, and if it does not, it can be easily adjusted.
  The pessary will be removed at 37 weeks of gestation, or before if any unexpected event occurs.
  Interventions: Device: Arabin Cervical Pessary

INTERVENTIONS:
Device: Arabin Cervical Pessary — The Arabin cervical pessary, which is CE-certified for preventing SPB (CE 0482 / EN ISO 13485: 2003 annex III of the council directive 93/42 EEC).
  It is a vaginal device which is used to treat pregnant women for preventing spontaneous preterm birth. This device can be easily placed around the uterine cervix without pain.
  Arms: Arabin Cervical Pessary

SUMMARY:
Placing a cervical pessary in severe twin-to-twin transfusion syndrome (TTTS) cases treated by fetoscopic laser coagulation (FLC) decreases the spontaneous preterm birth rate.

DETAILED DESCRIPTION:
Monochorionic (MC) twin pregnancies present with a high rate of fetal complications, most of them associated with the placental vascular anastomoses. Fetoscopic laser coagulation (FLC) is a surgical technique that allows minimally invasive access into the uterus and has emerged as a useful tool in the management of the most common and severe of these complications, twin to twin transfusion syndrome (TTTS). Even though, preterm birth remains a common cause of adverse outcome because TTTS is associated with a 29% risk of delivering before 28 weeks.

A short cervical length (CL), defined as a CL ≤ 25 mm, detected by transvaginal ultrasound is an independent risk factor for preterm birth in twin pregnancies but no effective treatment has been described to prevent it.

Although is usually accepted that in twin pregnancies cerclage may increase the risk of preterm birth, Salomon and co-workers, found that in cases of TTTS with a CL below the 5th percentile (15 mm) at the time of surgery, performing an emergency cerclage prolonged the pregnancy and allow for better outcome, But still preterm birth after FLC remains a big challenge, so new methods to prevent it must be investigated.

Previous studies in singletons and twins have shown that the use of cervical pessary significantly reduces the frequency of birth before 32 weeks and prolongs pregnancy. The advantage of using cervical pessary is that it is less invasive than cerclage and can be removed easily. That's the reason why pessaries could be considered an alternative, non invasive option to prevent preterm birth in cases of twin to twin transfusion syndrome (TTTS) treated by laser surgery.

ELIGIBILITY:
Inclusion Criteria:

* Monochorionic twin pregnancies with severe TTTS requiring intrauterine surgery
* Less than 26 weeks
* Minimal age of 18 years
* Informed consent signature

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* Cerclage prior to randomisation
* Uterine malformation
* Placenta previa
* Active vaginal bleeding at the moment of randomization
* Spontaneous rupture of membranes at the time of randomization
* Death of both twins after the surgery
* Monochorionic-monoamniotic twin pregnancy
* Silicone allergy
* Current participation in other RCT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Delivery before 32 weeks | Within the first 15 days after delivery
  Rate of delivery before 32 weeks

SECONDARY OUTCOMES:
Birth weight | Within the first 15 days after delivery
  Median weight (g) of the newborns at birth.
Fetal or neonatal death | Within the first 15 days after the death
  Rate of intrauterine demise or neonatal death during the first 24 hours.
Neonatal morbidity | 30 days after the discharge from the hospital
  Rate of major adverse neonatal outcomes before discharge from the hospital.
Significant maternal adverse events | Within 15 days after discharge from the hospital
  Rate of heavy bleeding (bleeding that requires a medical intervention), cervical tear (cervical rupture due to the pessary placement), and/or uterine rupture (rupture of the uterus due to contractions or surgery).
Physical or psychological intolerance to pessary | Within 15 days after discharge from hospital
  Discomfort or pain due to the pessary that makes daily life uncomfortable (number of cases).
Preterm birth before 37 weeks | Within 15 days after delivery
  Rate of delivery before 36+6 weeks
Rupture of membranes before 32 weeks | Within 15 days after delivery
  Rupture of amniotic membranes before 31+6 weeks
Hospitalisation for threatened preterm labour before 32 weeks | Within 15 days after delivery
  Requirement of hospitalisation due to preterm contractions that need medical treatment to try to stop them before 31+6 weeks (rate).
Time to birth | Within 15 days after delivery
Preterm birth before 34 weeks | Within 15 days after delivery
  rate of delivery before 33+6 weeks
Preterm birth before 30 weeks | Within 15 days after delivery
  rate of delivery before 29+6 weeks
Preterm birth before 28 weeks | Within 15 days after delivery
  rate of delivery before 27+6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena Carreras, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (4):
- UZ Leuven. Campus Gasthuisberg, Leuven, Belgium
- Germany (2):
  - Frauenklinik - Zentrum für Ultraschalldiagnostik und Pränatalmedizin Bürgerhospital und Clementine Kinderhospital gemeinnützige GmbH, Frankfurt
  - University Medical Center Eppendorf, Hamburg
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Carreras E, Arevalo S, Bello-Munoz JC, Goya M, Rodo C, Sanchez-Duran MA, Peiro JL, Cabero L. Arabin cervical pessary to prevent preterm birth in severe twin-to-twin transfusion syndrome treated by laser surgery. Prenat Diagn. 2012 Dec;32(12):1181-5. doi: 10.1002/pd.3982. Epub 2012 Oct 11. PMID 23055333
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493
- [Background] Goya M, Pratcorona L, Higueras T, Perez-Hoyos S, Carreras E, Cabero L. Sonographic cervical length measurement in pregnant women with a cervical pessary. Ultrasound Obstet Gynecol. 2011 Aug;38(2):205-9. doi: 10.1002/uog.8960. Epub 2011 Jul 18. PMID 21305638
- [Background] Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, Brons J, Duvekot H, Bijvank BN, Franssen M, Gaugler I, de Graaf I, Oudijk M, Papatsonis D, Pernet P, Porath M, Scheepers L, Sikkema M, Sporken J, Visser H, van Wijngaarden W, Woiski M, van Pampus M, Mol BW, Bekedam D. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicentre, open-label randomised controlled trial. Lancet. 2013 Oct 19;382(9901):1341-9. doi: 10.1016/S0140-6736(13)61408-7. Epub 2013 Aug 5. PMID 23924878
- [Derived] Rodo C, Maiz N, Arevalo S, Lewi L, Couck I, Hollwitz B, Kyvernitakis I, Carreras E, Hecher K. The Arabin cervical pessary for the prevention of preterm birth in twin-to-twin transfusion syndrome treated by fetoscopic laser coagulation: a multicenter randomized controlled trial. Am J Obstet Gynecol. 2024 Aug;231(2):252.e1-252.e11. doi: 10.1016/j.ajog.2023.11.1245. Epub 2023 Nov 29. PMID 38036166
- [Derived] Rodo C, Arevalo S, Lewi L, Couck I, Hollwitz B, Hecher K, Carreras E. Arabin cervical pessary for prevention of preterm birth in cases of twin-to-twin transfusion syndrome treated by fetoscopic LASER coagulation: the PECEP LASER randomised controlled trial. BMC Pregnancy Childbirth. 2017 Aug 1;17(1):256. doi: 10.1186/s12884-017-1435-0. PMID 28764674
- See also: Arabin Cervical Pessary — https://dr-arabin.de/product-category/products/obstetrics/?lang=en